CLINICAL TRIAL: NCT05322616
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Assess the Safety and Tolerability of JK07 in Subjects With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Single-Ascending Dose Study of JK07 in Subjects With HFpEF
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Salubris Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JK07.1.02
Record Dates: First submitted 2022-03-14; First posted 2022-04-12 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure; HFpHF; neuregulin-1
MeSH Terms: conditions — Heart Failure; Fibromatosis, Gingival, 2

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Single- Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matched placebo-solution
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JK07 (Active Comparator): Single dose of intravenous JK07 administered by intravenous infusion over 60 minutes.
  Interventions: Drug: JK07
- Matching Placebo (Placebo Comparator): Single dose of vehicle control administered by intravenous infusion over 60 minutes
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: JK07 — Recombinant fusion protein consisting of a fully humanized immunoglobulin G1 monoclonal antibody and an active polypeptide fragment of the human growth factor NRG-1
  Arms: JK07
Drug: Matching Placebo — Vehicle control
  Arms: Matching Placebo

SUMMARY:
A phase 1, randomized, double-blind, placebo-controlled single-ascending dose study to assess JK07 in adult subjects with heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
A phase 1, randomized, double-blind, placebo-controlled single-ascending dose study to assess the safety and tolerability of JK07 in subjects 18 to 85 years of age with heart failure with preserved ejection fraction (HFpEF) with left ventricular ejection fraction >=45%. Eligible subjects must have maintained an optimal heart failure medical regimen for at least 1 month prior to informed consent, other than for diuretics, and as much as clinically appropriate, remain on the treatment regimen throughout the course of the study.

Initially 5 dose escalation cohorts are planned with the option of expansion to 7 dose escalation cohorts. Eight subjects will be randomized in a 6:2 ratio of JK07:placebo in each cohort.

The initial dose and dose escalation parameters will be dependent on the JK07.1.01 study Only doses established as safe in Study JK07.1.01 will be evaluated in this study and the highest JK07 dose administered will not exceed the lower of the top dose evaluated in Study JK07.1.01 or 2.5 mg/kg without amending the protocol. Subjects will be observed in a hospital or similar setting from prior to study drug infusion to completion of study assessments on Day 1.

Subjects will undergo blood sampling for clinical laboratory evaluation, including glucose fingerstick, and biomarkers, electrocardiogram, 2-dimensional transthoracic echocardiography, quality of life assessment and a a 6-minute walking test. Follow-up assessments will be performed at Day 2, 7, 15, 28, 60, 90, and 180.

ELIGIBILITY:
Inclusion Criteria:

1. Stable New Yok Heart Association (NYHA) Class II or III HF diagnosis, evident at least 6 months prior to enrollment as confirmed by medical history.
2. Documented prior objective evidence of heart failure as shown by 1 or more of the following criteria:

   1. Previous hospitalization for heart failure with documented radiographic evidence of pulmonary congestion.
   2. Elevated left ventricular (LV) end-diastolic pressure or pulmonary capillary wedge pressure at rest (≥15 mm Hg) or with exercise (≥25 mm Hg).
   3. Elevated level of NT-proBNP (>400 pg/mL) or brain natriuretic peptide (BNP) (>200 pg/mL).
   4. Echocardiographic evidence of medial E/e' ratio ≥ 15 or Left Atrial Volume (LAV) >58 mL in male patients or >52 mL in female patients.
3. Adequate acoustic windows on screening resting TTE
4. Documented structural abnormality consistent with HFpEF confirmed at the screening visit by clearly interpretable echocardiography assessment.
5. Meets 1 or more of the following criteria at the initial screening measurement:

   1. A hs-cTnI >99th percentile
   2. NT-proBNP >300 pg/mL (if not in atrial fibrillation or atrial flutter) or >600 pg/mL (if in atrial fibrillation or atrial flutter), or if the screened participant is either of African descent or has a body mass index ≥30.0 kg/m2, a screening NT-proBNP >240 pg/mL (if not in atrial fibrillation or atrial flutter) or >480 pg/mL (if in atrial fibrillation or atrial flutter).
6. Body mass index (BMI) ≥18 kg/m2 and ≤45 kg/m2
7. Screening hemoglobin ≥9.0 g/dL, platelets ≥100x109 /mL, absolute neutrophil count (ANC) ≥1500/mL.
8. Sexually mature biological male subjects must agree to use a medically accepted method of contraception throughout the study and be willing and able to continue contraception until the end of the study (6-month time point).
9. Biological females of childbearing potential must present with a negative blood pregnancy test, must not be lactating, and must agree to employ adequate birth control measures for the duration of the study and be willing and able to continue contraception until the end of the study (6-month time point).
10. Subject is capable of giving signed informed consent.
11. Subject is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

Cardiac-Related

1. Participating in any other study and have received any other investigational drug within 30 days prior to screening or 5-half-lives, whichever is longer, or any other investigational implanted device within 30 days prior to screening, or are taking part in a nonmedication study which, in the opinion of the Investigator, would interfere with study compliance or outcome assessments.
2. Any past participation in a study that has investigated the NRG-1 pathway (e.g., Neucardin, cimaglermin).
3. Has a prior diagnosis of hypertrophic cardiomyopathy or a known infiltrative or storage disorder causing HFpEF and/or cardiac hypertrophy, such as amyloidosis, Fabry disease, or Noonan syndrome with LV hypertrophy or a positive serum immunofixation result.
4. Has a history of syncope within the last 6 months or sustained ventricular tachycardia with exercise within the past 6 months.
5. Has persistent or permanent atrial fibrillation and is not therapeutically anticoagulated for at least the 4 weeks prior to the initial screening visit or is not adequately rate controlled within 6 months prior to informed consent according to investigator discretion.
6. Has known moderate or severe aortic valve stenosis, hemodynamically significant mitral stenosis, or severe mitral or tricuspid regurgitation at informed consent.
7. Has severe chronic obstructive pulmonary disease, or other severe pulmonary disease, requiring home oxygen, chronic nebulizer therapy, chronic oral steroid therapy or hospitalized for pulmonary decompensation within 12 months of informed consent.
8. Diagnosed with medically documented acute coronary syndrome within 3 months of screening or a medically documented acute myocardial infarction within 6 months of screening.
9. Cardiac surgery, coronary artery revascularization, percutaneous coronary intervention, or valvuloplasty within 3 months prior to screening.
10. Any subject who has received an indication for coronary revascularization within 3 months prior to screening.
11. Any of the following confirmed by duplicate seated determinations on at least 3 consecutive readings (in clinic/office) following informed consent and prior to randomization:

    1. Systolic blood pressure (SBP) ≥160 mmHg and/or diastolic blood pressure (DBP) >100 mmHg
    2. Sustained SBP <90 mmHg and/or DBP <40 mmHg and/or symptomatic hypotension
    3. Sustained resting heart rate (HR) <50 or ≥100 bpm or >110 bpm if chronic AF at Screening (Visit 1) or prior to randomization for >15 minutes in two episodes separated by one hour of observation
12. Cerebrovascular accident or hospitalizations for cardiovascular (CV) causes other than routine percutaneous procedures (such as device, battery, generator changes or pacemaker lead insertion/replacement), including HF, chest pain, stroke, transient ischemic attack, or arrhythmias within 3 months prior to screening.
13. Symptomatic carotid stenosis or transient ischemic attack or stroke within 60 days prior to informed consent.
14. Has a history of resuscitated sudden cardiac arrest or a known history of appropriate implantable cardioverter-defibrillator (ICD) discharge for life-threatening ventricular arrhythmia. (Note: history of anti-tachycardia pacing (ATP) is allowed.)
15. Subjects at screening have an abnormal or clinically significant 12-lead ECG abnormality, that, in the opinion of the Investigator, would affect efficacy or safety evaluation or place the subject at risk.
16. History or evidence of clinically significant arrhythmias uncontrolled by drug therapy or use of an implantable defibrillator, long QT syndrome, or evidence of QT prolongation with QTcF >450 ms for males or QTcF >470 ms for females during screening and/or prior to randomization.

    Non-Cardiac Co-Morbidity
17. Clinically significant renal dysfunction as measured by the estimated glomerular filtration rate of <45 mL/min/1.73m2 as calculated by local laboratory standards (Cockcroft-Gault equation for estimation of creatinine clearance [CrCl] [Cockcroft and Gault 1976]) at screening, or a clinically significant change in renal function between screening and baseline.
18. Clinically significant liver dysfunction as measured by: alanine aminotransferase (ALT) >2.0 × the upper limit of normal (ULN), alkaline phosphatase > 2.0 × ULN, aspartate aminotransferase (AST) >2.0 × ULN, or gamma glutamyl transferase (GGT) >2.0 × ULN or serum bilirubin ≥ 1.5 × ULN at screening, or a clinically significant change in liver function between screening and baseline.
19. Subjects with alteration of the coagulation panel (international normalized ratio [INR]) and/or prothrombin time (PT) ≥1.5 × the ULN; activated partial thromboplastin time (aPTT) ≥1.5 × ULN, or serum albumin ≤3 gm/dL. For subjects on warfarin or other anticoagulants, an INR (or PT) considered by the Principal Investigator as therapeutically appropriate will be allowed.
20. Any subject who by Investigator's judgement, has a significant hematuria or proteinuria at screening.
21. Concurrent treatment with Class Ia or III antiarrhythmic drugs if the dosage has been adjusted within 2 months prior to informed consent.
22. Positive screening for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies.
23. Known history of or active alcohol abuse (no more than 14 units/week for males or 7 units/week for females) or use of illicit drugs within 1 year prior to randomization (excluding recreational use of marijuana or cannabidiol [CBD]-based products).
24. Other medical or psychiatric condition that, in the opinion of the Investigator, would preclude obtaining voluntary consent/assent or would confound the secondary objectives of study.
25. A history of pathologically confirmed malignancy of any type or any pathologically confirmed pre-malignant condition (e.g., ductal carcinoma in situ, colonic polyp with premalignant diagnosis, or cervical atypia). All subjects are to undergo cancer screening following study enrollment in accordance with American Cancer Society Guidelines (See Appendix 1).
26. Pregnant or lactating at screening.
27. Subjects with clinically significant or poorly controlled disease including, but not limited to, endocrine (including diabetes and thyroid) disease, pulmonary (requires home oxygen, inhalants, steroids >10 mg prednisone equivalent or 2x baseline physiologic steroid replacement, primary pulmonary hypertension, history of pulmonary emboli), neurological or psychiatric (even mild), GI, hematological, urological, immunological, ophthalmic, or orthopedic diseases as determined by the Investigator.
28. Any major surgical procedure within 1 month prior to screening or planned surgical procedure during the study period.
29. Subjects who are not non-smokers or light smokers (no more than 5 cigarettes per day) and who cannot abstain from smoking from 2 weeks prior to the administration of IP through the end of the study.
30. Subjects with orthopedic impairment which would prohibit credible or adequate assessment of 6MWT.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Safety Assessment | Screening to Day 28
  Incidence and severity of treatment-emergent adverse events (safety and tolerability) by assessment of physical exams, injection site, vital signs and clinical laboratory tests.

OTHER OUTCOMES:
Natriuretic peptide | Screening to Day 180
  Change in brain natriuretic peptide (BNP) and N-terminal pro-brain natriuretic peptide (NTpro-BNP) change from baseline
Quality of Life - Kansas City Cardiomyopathy Questionnaire (KCCQ) | Screening to Day 180
  Change from baseline in the Clinical Summary Score of the KCCQ, a 23-item self-administered questionnaire that measures the patient's perception of their health status including symptoms of heart failure (eg., shortness of breath, fatigue, edema) and impact on physical and social function
6-Minute Walking Test (6MWT) | Screening to Day 180
  Change from baseline in the 6MWT
Two-dimensional Transthoracic Echocardiography (2D-TTE) | Screening to Day 180
  Change from baseline to each assessment time point for 2D-TTE indices including but not limited to change in Echocardiographic evidence of medial E/e' ratio, Left Atrial Volume (LAV) in mL, LAV index in mL/m2, Left Atrial Area (LAA) in cm2

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (7):
  - Stanford University Medical Center, Stanford, California
  - Harvard Medical School/Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No